CLINICAL TRIAL: NCT06114329
Title: A Phase II, Open-label Study to Evaluate the Safety, Pharmacodynamics, Pharmacokinetics, and Efficacy in Males With Classic Fabry Disease Who Have Never Received Any Treatment
Brief Title: Study of the Safety and Biologic Activity of AL01211 in Treatment Naive Males With Classic Fabry Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AceLink Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AL01211-202
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2023-11

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AL01211 30 mg, once daily (Experimental): 9 subjects will first be enrolled in this arm, receiving 30 mg AL01211 treatment, once daily
  Interventions: Drug: AL01211
- AL01211 60 mg, once daily (Experimental): After enrolling into 30 mg arm is completed and preliminary data show good safety, 9 subjects will be enrolled in this arm, receiving 60 mg AL01211 treatment, once daily
  Interventions: Drug: AL01211

INTERVENTIONS:
Drug: AL01211 — AL01211 is a novel, proprietary, selective GCS inhibitor with high potency against GCS with limited off target activity.

SUMMARY:
This is a Phase II, open-label study designed to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of AL01211 in male subjects with classic Fabry disease who have never received any treatment (eg. ERT or chaperone therapy). Eligible subjects will receive 182 days (26 weeks) of study treatment as the primary study period followed by an extension period. The total study duration for a subject is up to at most 2 years including the primary period of 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with classic Fabry mutations with between 18 and 60 years of age, inclusive, at screening.
* Have never received any Fabry disease-specific treatment (eg. ERT, chaperone therapy).
* Signed and dated informed consent prior to any study mandated procedure.
* Confirmed diagnosis of Fabry disease as documented by the presence of a Fabry genetic variant of known significance and documented (within 10 years prior to study entry) leukocyte αGAL activity of <4 nmol/hr/mg or plasma αGAL activity of <1.5 nmol/hr/mL. If the genetic variant is not known or available, genetic test will be done to document the genetic variation after obtaining the patient's informed consent. If documented leukocyte or plasma αGAL activity is unavailable, the subject must consent to plasma αGAL activity screening.
* eGFR ≥50 mL/min/1.73 m2 by CKD-EPI Creatinine-Cystatin Equation (2021) at the screening visit.
* Subject agrees to comply with all procedural requirements as presented in the protocol, including participation in observational period which extends beyond the planned 52-week treatment duration of the study and 1 month follow-up visit.
* For subjects receiving renin-angiotensin-aldosterone system (RAAS) inhibitors/blockers (ACEIs, ARBs, aldosterone receptor antagonists) or sodium-glucose cotransporter-2 (SGLT2) inhibitors, the dose should be stable (ie, prescribed dose and frequency) for at least the immediate 3 months prior to screening.
* Symptom or clinical finding of ≥1 of the characteristic features of Fabry disease, such as, but not limited to, neuropathic pain, symptoms of gastrointestinal, renal, or cardiac dysfunction.
* Willing to undergo opthalmological examination with photodocumentation at baseline and at specified times during the study.
* Plasma Lyso GL3 ≥25 ng/mL.

Exclusion Criteria:

* Subject on regular dialysis for the treatment of chronic kidney disease or has undergone a kidney transplant.
* Clinically significant abnormal liver function judged by the investigator, including but not limited to serum total bilirubin > 1.5 the upper limit of normal [ULN], serum alanine aminotransferase > 2 times the ULN, or aspartate aminotransferase >2 times the ULN).
* Scheduled in-patient hospitalization, including elective surgery, during the study.
* A positive result on any of the following tests: hepatitis B surface antigen (HBsAg) (If HBsAg is positive, hepatitis B virus DNA needs to be tested, and the copy number >ULN), antihepatitis C virus antibodies, anti-human immunodeficiency virus 1 and 2 antibodies.
* A cortical cataract (COR) >one quarter of the lens circumference (Grade COR-2) or a posterior subcapsular cataract (PSC) with about 30% opacity (Grade PSC-2), according to World Health Organization grading. Subjects with nuclear cataracts are not excluded.
* Currently receiving, or has received within the past month, potentially cataractogenic medications, including a chronic regimen (more frequently than once every 2 weeks) of any route of corticosteroids (limited to medium and high-potency topical steroids; intranasal steroids are acceptable) or any medication that may cause cataracts (such as phenothiazines and miotics, amiodarone, allopurinol and phenytoin) according to the Prescribing Information.
* Male subjects with partners of child-bearing potential who do not agree to use a medically accepted, highly eﬀective method of contraception during the study until 3 months after the last administration of study drug. Male subjects must be willing to withhold from any sperm donation during the study and up to 3 months after the last dose of study treatment.
* Presence of any medical, emotional, behavioral, or psychological condition that, in the judgment of the investigator, would interfere with the subject's compliance with the requirements of the study or interpretation of the results.
* Prior participation in a study involving an investigational drug within 90 days since the end of the study or within 5 half lives since the last dose of investigational drug, whichever is longer.
* Unwilling to comply with the requirements of the protocol.
* Known and documented cardiovascular event (eg, myocardial infarction, unstable angina), cerebrovascular event (eg, stroke, transient ischemic attack), or clinically significant unstable cardiac disease (eg, uncontrolled symptomatic arrhythmia or congestive heart failure of New York Heart Association Class III or IV) in the 6 months prior to screening.
* Any cardiac disease that could mimic Fabry disease or confound cardiac measurement, such as (non-Fabry related) hypertrophic cardiomyopathy or the presence of a pacemaker or implantable cardioverter/defibrillator; any contraindications to MRI measurement (eg, cerebral aneurysm clips).
* History of acute kidney injury in the 12 months prior to screening, including specific kidney diseases (eg, acute interstitial nephritis, acute glomerular and vasculitic renal diseases), nonspecific conditions (eg, ischemia and toxic injury), and extrarenal pathology (eg, prerenal azotemia and acute postrenal obstructive nephropathy).
* Subjects received herbal medicines within 14 days prior to screening.
* The participant had received strong or moderate inducers or inhibitors of Cytochrome P450 3A4 (CYP3A4) within 14 days prior to enrollment or within 5 times the elimination half-life or PD half-life of the medication, whichever is longer; Ingested grapefruit, grapefruit juice, or grapefruit products within 72 hours prior to initial administration, or were unwilling to avoid grapefruit, grapefruit juice, or grapefruit products during treatment.
* Any other situations that the investigator considers unsuitable for the patient to participate in this study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | 104 weeks
  Number of subjects with TEAEs will be evaluated. AEs will be coded by using the current version of the Medical Dictionary for Regulatory Activities and summarized by system organ class, preferred term, and dose level for the number and percent of AEs reported, the number of subjects reporting each AE, and the number of subjects with any AE.

SECONDARY OUTCOMES:
The pharmacodynamics of AL01211 by measuring plasma GL1 level | Baseline, weeks 2, 4, 8, 13, 26, 52, 104
  Plasma level of GL1 will be determined by Liquid Chromatography with tandem mass spectrometry (LC-MS-MS).
The pharmacodynamics of AL01211 by measuring plasma GL3 level | Baseline, weeks 2, 4, 8, 13, 26, 52, 104
  Plasma levels of GL3 will be determined by Liquid Chromatography with tandem mass spectrometry (LC-MS-MS).
The pharmacodynamics of AL01211 by measuring plasma lyso globotriaosylceramide (Lyso GL3) level | Baseline, weeks 2, 4, 8, 13, 26, 52, 104
  Plasma levels of Lyso-GL3 will be determined by Liquid Chromatography with tandem mass spectrometry (LC-MS-MS).
The pharmacodynamics of AL01211 by measuring urine GL3 level | Baseline, weeks 4, 13, 26, 52, 104
  Urine levels of GL3 will be determined by Liquid Chromatography with tandem mass spectrometry (LC-MS-MS).
The pharmacodynamics of AL01211 by measuring urine lyso globotriaosylceramide (Lyso GL3) level | Baseline, weeks 4, 13, 26, 52, 104
  Urine levels of Lyso-GL3 will be determined by Liquid Chromatography with tandem mass spectrometry (LC-MS-MS).
The pharmacokinetics of AL01211 in plasma | Weeks 1, 2, 4, 8, 13, 26, 52, 104
  Plasma samples will be collected, and AL01211 plasma concentrations will be measured with Liquid Chromatography with tandem mass spectrometry (LC-MS/MS).
The pharmacokinetics of AL01211 in urine | weeks 1 and 13
  Urine samples will be collected, and AL01211 urine concentrations will be measured with Liquid Chromatography with tandem mass spectrometry (LC-MS/MS).
The effect of AL01211 on renal function: eGFR | 104 weeks
  Change from Baseline in estimated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine-Cystatin Equation (2021) at Weeks 2, 4, 8, 13, 26, 52, 104.
The effect of AL01211 on renal function: UPCR | 104 weeks
  Change from Baseline in urine protein/creatinine ratio (UPCR) at Weeks 13, 26, 52, 104.
The effect of AL01211 on renal function: UACR | 104 weeks
  Change from Baseline in urine albumin/creatinine ratio (UACR) at Weeks 13, 26, 52, 104.
The effect of AL01211 on cardiac function: MRI±gadolinium | 104 weeks
  Change from Baseline in MRI±gadolinium measurements at Weeks 26, 52, 104.
The effect of AL01211 on cardiac function: troponin T | 104 weeks
  Change from Baseline in plasma troponin T level at Weeks 2, 4, 8, 13, 26, 52 and 104.
The effect of AL01211 on symptoms of neuropathic pain: BPI-SF | 104 weeks
  Change from Baseline in Brief Pain Inventory-Short Form (BPI-SF) at Weeks 4, 8, 13, 26, 52, 104.
The effect of AL01211 on symptoms of neuropathic pain: average weekly pain severity during Fabry crises | 104 weeks
  Change from Baseline in average weekly pain severity during Fabry crises (episodic pain attacks) as assessed by an 11-point Numeric Rating Scale (NRS) at Weeks 4, 8, 13, 26, 52, 104.
The effect of AL01211 on symptoms of neuropathic pain: weekly frequency of Fabry crises | 104 weeks
  Change from Baseline in weekly frequency of Fabry crises (episodic pain attacks) at Weeks 4, 8, 13, 26, 52, 104.
The effect of AL01211 on symptoms of neuropathic pain: weekly frequency of use of pain medication | 104 weeks
  Change from Baseline in weekly frequency of use of pain medication at Weeks 4, 8, 13, 26, 52, 104.
The effect of AL01211 on symptoms of gastrointestinal disturbance | 104 weeks
  Change from Baseline in average weekly gastrointestinal symptom diary up to at Weeks 4, 8, 13, 26, 52, 104.
The pharmacodynamics of AL01211 by measuring GL3 inclusion in kidney biopsies | Baseline, weeks 52, and 104
  Change from baseline in histological scoring of the number of GL-3 inclusions per kidney interstitial capillary (KIC) at Week 52 and 104. (optional)
The effect of AL01211 on quality of life: EQ-5D-5L | 104 weeks
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Change from Baseline in EQ-5D-5L at Weeks 13, 26, 52 and 104 will be assessed.
The effect of AL01211 on overall disease burden | 104 weeks
  Fabry Outcome Survey Mainz Severity Score Index (FOS-MSSI) is a tool for clinicians to evaluate the severity and progression of Fabry disease in adult patients. A higher score on FOS-MSSI means a higher disease burden. It will be assessed at Weeks 13, 26, 52 and 104
The effect of AL01211 on clinician reported global impression of severity of disease | 104 weeks
  Change from Baseline in Clinical Global Impression of Severity (CGI-S) score at Weeks 4, 8, 13, 26, 52 and 104. A higher score (from 0 to 3) means a greater severity.
The effect of AL01211 on clinician reported global impression of change of disease | 104 weeks
  Change from Baseline in Clinical Global Impression of Change (CGI-C) score assessed at Weeks 4, 8, 13, 26, 52 and 104. A higher score (from 1 to 5) means a greater overall worsening of symptoms.
The effect of AL01211 on patient reported global impression of severity of disease | 104 weeks
  Change from Baseline in Patient Global Impression of Severity (PGI-S) score assessed at Weeks 4, 8, 13, 26, 52 and 104. A higher score (from 0 to 3) means a greater severity.
The effect of AL01211 on patient reported global impression of change of disease | 104 weeks
  Change from Baseline in Patient Global Impression of Change (PGI-C) score assessed at Weeks 4, 8, 13, 26, 52 and 104. A higher score (from 1 to 5) means a greater overall worsening of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Chen, Dr., Principal Investigator — Ruijin Hospital
Locations (6):
- China (6):
  - The First Affiliated Hospital of Sun Yat sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing
  - Ruijin Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai